CLINICAL TRIAL: NCT03576443
Title: A Phase II Trial of Idelalisib in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Trial of Idelalisib in Patients With Relapsed Diffuse Large B-cell Lymphoma
Acronym: ILIAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-LBC-07
Record Dates: First submitted 2018-04-30; First posted 2018-07-03 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Idelalisib 150 mg x 2 p o, until progression
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg x 2 p o

SUMMARY:
Based on the high response rate in heavily pretreated patients with indolent B-cell lymphomas, among which it is likely that many have undetected transformed disease, the investigators hypothesize that idelalisib may also be active in relapsed DLBCL, particularly of the GCB subtype. Possibly, the efficacy may be related to the presence of specific mutations within the B-cell receptor pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) , including transformed low grade lymphoma, with either:

   1. Refractory disease: defined as disease progression while receiving their most recent prior cytotoxic chemotherapy (single-agent immunotherapy as maintenance is not considered cytotoxic therapy).
   2. Persistent disease: defined as stable disease or partial response at the completion of their most recent prior cytotoxic chemotherapy.
   3. Relapsed/recurrent disease: defined as complete response at the end of their most recent prior cytotoxic chemotherapy with subsequent relapse or disease recurrence.
3. Subjects must have received prior rituximab and may have received up to 5 prior regimens containing cytotoxic chemotherapies.
4. Subjects must not be candidates for high-dose chemotherapy with autologous stem cell support (ASCT), due to one or more of the following factors: relapse after high dose chemotherapy, age, comorbid disease, performance status, or persisting toxicities from prior chemotherapy.
5. Absolute neutrophil count (ANC) >1.0 x 109/L, unless related to bone marrow infiltration.
6. At least 1 measurable disease lesion that is >1.0 cm in 2 perpendicular dimensions, with the product diameter >2.25 cm2 by computed tomography (CT) or magnetic resonance imaging (MRI).
7. Negative serum pregnancy test within 1 week before first treatment if the subject is a woman of childbearing potential. The use of highly-effective contraception methods* are required during the study for women of child-bearing potential. Due to the toxicity of idelalisib, women who will use a hormonal contraceptive must in addition also use a barrier method, since it is currently unknown whether idelalisib may reduce the effectiveness of hormonal contraceptives. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
8. WHO performance status 0 - 3.
9. Written informed consent.

Exclusion Criteria:

1. Prior allogeneic hematopoietic stem cell transplant (HSCT).
2. Prior treatment with PI3K inhibitors.
3. Serum total bilirubin ≥ 1.5 x ULN (unless elevated due to Gilbert's syndrome).
4. Serum ALT and AST ˃ 2.5 x ULN.
5. Estimated Creatinine Clearance < 10 ml/min.
6. Known seropositivity for human immunodeficiency virus (HIV).
7. Known history of drug induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver or portal hypertension.
8. Known history of drug induced pneumonitis.
9. On-going inflammatory bowel disease.
10. Evidence of serious active infection (eg, requiring an intravenous [IV] antibiotic, antiviral, or antifungal agent), or subjects with a recent history of deep tissue infections such as fascitis or osteomyelitis.
11. Chemotherapy, cancer immunosuppressive therapy, growth factors (except erythropoietin), or investigational drugs/devices <10 days before first dose of investigational product in this study. Subjects receiving high doses of corticosteroids must have been tapered to a stable dose at least 7 days before the first dose of investigational product.
12. Pregnant or breastfeeding women.
13. Symptomatic central nervous system (CNS) NHL; a lumbar puncture is not required unless CNS involvement with NHL is clinically suspected.
14. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition).
15. Concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix. Subjects with previous malignancies are eligible provided that they have been disease free for >2 years.
16. Previous myocardial infarction or pulmonary hypertension <6 months before first dose of investigational product.
17. History of clinically significant ventricular arrhythmia, prolonged QTc interval or unexplained syncope.
18. Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate for GCB DLBCL | at time of progression, up to 112 weeks from start of treatment
  Overall response rate (ORR) for GCB DLBCL

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, Principal Investigator — Department of Oncology Skåne University Hospital
Locations (6):
- Denmark (2):
  - Aarhus University Hospital, Aarhus C
  - Odense University Hospital, Odense
- Sweden (4):
  - Halmstad County Hospital, Halmstad
  - Linkoping University Hospital, Linköping
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No